CLINICAL TRIAL: NCT01338857
Title: Phase II Study of Sorafenib in Children and Young Adults With Recurrent or Progressive Low-Grade Astrocytomas
Brief Title: Sorafenib in Children and Young Adults With Recurrent or Progressive Low-Grade Astrocytomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sorafenib ineffective for tx of recurrent or progressive PLGA
Sponsor: NYU Langone Health (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-00561
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2016-12

CONDITIONS: neurofibromatosis1 (NF1); Recurrent or Progressive Optic Pathway Gliomas (OPG); Recurrent or Progressive Low-grade Glioma
Keywords: neurofibromatosis1 (NF1); Recurrent or progressive optic pathway gliomas (OPG); Recurrent or progressive low-grade glioma; sorafenib; low-grade astrocytoma
MeSH Terms: conditions — Recurrence | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Nexavar) (Experimental): Sorafenib will be administered orally BID (approximately every 12 hours). Grapefruit juice is not allowed while taking sorafenib. A cycle of therapy is considered to be 28 days and there is no interruption between cycles. Patients may receive up to a total of 12 cycles provided that no off-protocol or off-study criteria are met.
  Interventions: Drug: Sorafenib (Nexavar)

INTERVENTIONS:
Drug: Sorafenib (Nexavar) — Sorafenib (in tablet form) will be administered orally BID (approximately every 12 hours). Grapefruit juice is not allowed while taking sorafenib. A cycle of therapy is considered to be 28 days and there is no interruption between cycles. Patients may receive up to a total of 12 cycles provided that no off-protocol or off-study criteria are met.
  Children/adolescents (< 18 years of age, non-NF1): 200 mg/m2/dose PO twice daily (rounded to the nearest 50 mg increment as per Section 4.1) to a maximum of 400 mg PO twice daily
  Adults (greater than or equal to 18 years of age, non-NF1): 400 mg PO twice daily
  NF1 patients (regardless of age): 80 mg/m2/dose PO twice daily (rounded to the nearest 50 mg increment as per Section 4.1) to a maximum of 150 mg PO twice daily

SUMMARY:
The purpose of this study is to determine if a drug called sorafenib can shrink LGA tumors (low-grade astrocytomas) in children and adults. Previous research has given us a better understanding of this type of tumor by studying the genetic "make-up" of LGAs. From this research, the investigators found that a drug called sorafenib may stop the growth of tumor cells by blocking some of the molecules needed for cell growth and by blocking blood flow to the tumor. This trial is studying how well sorafenib works in treating patients with LGAs, and how the effects relate to the specific genetic "make-up" of your particular tumor. This testing of your tumor's genetic make-up is optional and requires available tumor tissue for testing. In summary, the aims of this study are: To see if sorafenib can shrink LGAs; how well sorafenib is tolerated in patients with LGAs; and, how the effects of sorafenib relate to the genetic make-up of individual LGAs (Optional Study)

DETAILED DESCRIPTION:
Novel therapies are urgently needed for children with relapsed LGA who are not surgical candidates and/or have exhausted standard chemotherapy approaches. Although a vast number of "molecular targeted" agents have been developed over the past decade for the treatment of cancer, none have been evaluated for the treatment of LGAs. Recently, genetic alterations resulting in oncogenic BRAF have been identified to be highly prevalent in LGAs, providing a rational target for therapeutic intervention.

The aims of this clinical trial are to estimate the efficacy, as well as safety and tolerability of sorafenib, a RAF and tyrosine kinase receptor inhibitor, in the treatment of pediatric patients with recurrent LGA. Sorafenib targets several pathways that, based on preliminary data from us and others, are likely contributing to the growth of LGAs: oncogenic BRAF, which is present in the majority of grade I LGAs and VEGFR2 and PDGFR, which are well-described mediators of tumor angiogenesis. Since sorafenib inhibits a number of additional kinases whose role in LGA growth has not yet been explored, it is possible that inhibition of pathways other than the primary targets may result in additional anti-tumor effects of sorafenib in LGA. Although the investigators hypothesize that LGAs with oncogenic BRAF should be most sensitive to sorafenib, the additional targets of sorafenib may also result in significant anti-tumor effects in LGAs with wild-type BRAF. Therefore, the investigators propose to evaluate the efficacy of sorafenib in children with LGAs in a translational clinical trial, stratified by BRAF status and tumor grade.

The investigators expect to learn the following from this clinical translational trial:

* The anti-tumor activity of sorafenib in pediatric LGAs
* The safety and tolerability of sorafenib in pediatric patients with LGAs
* The association of molecular target expression, e.g. oncogenic BRAF, with response rates

The investigators will use the results of the clinical translational trial to determine if sorafenib warrants further clinical study in pediatric LGAs. If the investigators find associations between molecular target expression and response, further studies may be limited to or focus on patients whose tumors have specific molecular features, such as oncogenic BRAF. Sorafenib has also shown promise in combination with classic chemotherapy and can be given together with carboplatin, which is one of the most active agents in LGAs. Therefore, possible synergy between sorafenib and traditional chemotherapy used in the treatment of LGAs, such as carboplatin, could be explored in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age: greater than or equal to 2 years of age
* Patients with neurofibromatosis-1 (NF1) are eligible
* Recurrent/progressive optic pathway gliomas (OPG) by MRI criteria, after standard therapy - histologic confirmation not required OR Histologically confirmed, radiographically recurrent or progressive low-grade glioma (WHO grade I or II) by MRI criteria, after standard therapy.
* Karnofsky performance status (PS) 60-100% (greater than or equal to 16 years of age) OR Lansky PS 60-100% (< 16 years of age)
* Absolute neutrophil count ≥ 1,000/mm³ (unsupported)
* Platelet count ≥ 75,000/mm³ (unsupported)
* Normal PT, PTT, and INR (for patients on prophylactic anticoagulation only)
* Diastolic blood pressure (DBP) ≤ the 95th percentile for age and gender and not currently receiving medication for the treatment of hypertension.
* Adequate pulmonary function, defined as: no evidence of dyspnea at rest, no exercise intolerance, and pulse oximetry > 94% if termination is clinically indicated.
* Not received myelosuppressive chemotherapy or treatment with biologicals or monoclonal antibodies within 4 weeks of enrollment onto this study (6 weeks if prior nitrosurea)
* At least 7 days since the completion of therapy with a hematopoietic growth factor and at least 14 days from the last administration of PEGylated GCSF (Neulasta®)
* If prior radiation therapy, ≥ 6 months must have elapsed since the last fraction for craniospinal therapy and ≥ 3 months for focal radiotherapy including radiosurgery.
* If prior surgery, ≥ 8 weeks must have elapsed since (≥ 4 weeks for minor surgery/procedures including central line placement)
* Steroids are allowed for progressive symptoms but patient must be on a stable or decreasing dose for at least 1 week prior to study entry
* Any neurologic deficits must be stable for ≥ 1 week

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness, including overt hepatic or renal disease, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
* Baseline hypertension greater than grade 1.
* Prior treatment with sorafenib
* Other concurrent investigational drugs
* Other concurrent anticancer agents or therapies, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy
* Concurrent therapeutic anticoagulation. Prophylactic anticoagulation (i.e. low dose heparin) of venous or arterial access devices is allowed.
* Concurrent administration of any of cytochrome P450 enzyme-inducing agents, including grapefruit juice and drugs listed under Section 9.7.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event
* Any other hemorrhage/bleeding event
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of unresolved bleeding diathesis or coagulopathy.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Known or suspected allergy to sorafenib.
* Any malabsorption problem.
* Patients with history of any prior CNS bleeding.
* Patients with any non-healed wounds.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias A Karajannis, MD, Principal Investigator — NYU
Locations (1):
- New York University Stephen D. Hassenfeld Children's Center for Cancer & Blood Disorders, New York, New York, United States

REFERENCES:
- [Derived] Legault G, Kieran MW, Scott RM, Chordas C, Milla SS, Karajannis MA. Recurrent ascites in a patient with low-grade astrocytoma and ventriculo-peritoneal shunt treated with the multikinase inhibitor sorafenib. J Pediatr Hematol Oncol. 2014 Nov;36(8):e533-5. doi: 10.1097/MPH.0000000000000094. PMID 24351969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened to recruitment 4/13/2011 and ended on 4/24/2012. Recruitment took place at the NYU Hassenfeld Children's Center outpatient clinic.
Pre-assignment Details: Participants were not excluded from the trial before assignment to groups. Treatment was based on age and diagnosis of neurofibromatosis type I.
Groups:
- Sorafenib (Nexavar): Sorafenib will be administered orally BID (approximately every 12 hours). A cycle is 28 days w/o interruption between cycles. Patients may receive up to a total of 12 cycles provided that no off-protocol or off-study criteria are met.
  Children/adolescents (< 18 years of age, non-NF1): 200 mg/m2/dose PO twice daily (rounded to the nearest 50 mg increment) to a maximum of 400 mg PO twice daily
  Adults (greater than or equal to 18 years of age, non-NF1): 400 mg PO twice daily
  NF1 patients: 80mg/m2/dose PO 2x daily to max of 150mg PO 2x daily.
Period: Overall Study
Arm/Group | Sorafenib (Nexavar)
Started | 12
Completed | 1
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib (Nexavar)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.25 (3)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Response Rate to Sorafenib
Description: To estimate the objective response rates to sorafenib in children and young adults with low-grade astrocytomas, including optic pathway gliomas.
Time Frame: one year
Population: Study terminated and 1/12 participants completed and data was analyzed
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar)
Number analyzed (Participants) | 1
participants | 1

2. Primary Outcome: Objective Response Rates
Description: Determination of tumor response (CR, PR, SD) will be defined based on the comparison of the baseline MRI performed at study entry to the subsequent MRI which demonstrated best response. PR will be defined by a >15% decrease in tumor volume, as measured by 3D volumetric analysis.
Time Frame: MRIs performed after every 3rd 28-day cycle and off-study
Population: Study terminated and 1/12 participants completed and data was analyzed
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar)
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Arm/Group | Sorafenib (Nexavar)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (Nexavar) (N=12)
ALT increase (Investigations) | 5 (6)
anal hemorrhage (Gastrointestinal disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 1 (1)
ascites (Gastrointestinal disorders) | 1 (1)
AST elevation (Investigations) | 8 (9)
blood in stool (Gastrointestinal disorders) | 1 (2)
cold symptoms (runny nose) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
conjunctivitis (Eye disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
decreased appetite (Metabolism and nutrition disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 7 (8)
dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
emesis (Gastrointestinal disorders) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 2 (5)
eye pain (Eye disorders) | 1 (1)
fatigue (General disorders) | 4 (5)
fever (General disorders) | 1 (1)
flushing (facial) (Vascular disorders) | 2 (2)
gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
GGT (Investigations) | 1 (2)
hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4 (7)
headache (Nervous system disorders) | 3 (3)
hyperglycemia (Metabolism and nutrition disorders) | 4 (9)
hyperkeratotic eruptions (Skin and subcutaneous tissue disorders) | 1 (4)
hypernatremia (Metabolism and nutrition disorders) | 2 (2)
hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
hypertension (Vascular disorders) | 2 (2)
hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
hypokalemia (Metabolism and nutrition disorders) | 3 (5)
hyponatremia (Metabolism and nutrition disorders) | 5 (10)
hypophosphatemia (Metabolism and nutrition disorders) | 5 (6)
hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
intracranial pressure (Nervous system disorders) | 1 (1)
lethargy (Nervous system disorders) | 2 (2)
lymphocyte count decreased (Investigations) | 2 (2)
lymphopenia (Investigations) | 1 (1)
mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
muscle weakness-right sided (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
neutrophil count decreased (Investigations) | 3 (3)
papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1)
platelet count decreased (Investigations) | 2 (2)
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
ptosis (CN III) (Eye disorders) | 1 (1)
PTT (Investigations) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 10 (13)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
skin ulceration (nasal) (Skin and subcutaneous tissue disorders) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
tooth pain (Gastrointestinal disorders) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
UTI (Infections and infestations) | 1 (1)
vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 5 (6)
watery and itchy eyes (Eye disorders) | 1 (1)
white blood cell decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No